CLINICAL TRIAL: NCT03595007
Title: The Heroes Circle Opioid Project
Acronym: HCOP
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Other Study IDs: HCOP
Record Dates: First submitted 2018-06-19; First posted 2018-07-23 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Phase 1
  Interventions: Behavioral: Kids Kicking Cancer program
- Phase 2
  Interventions: Behavioral: Kids Kicking Cancer program
- Phase 3
  Interventions: Behavioral: Kids Kicking Cancer program

INTERVENTIONS:
Behavioral: Kids Kicking Cancer program — Individual instruction on how to lower stress and life challenges. Patient and martial artist will work together to identify obstacles that interfere with methadone goal reduction. Training will include learning certain martial arts rituals and breathing techniques. Patients will receive audio meditations for smart phone devices and regular reminders to practice. Each weekly meeting will be supplemented by 3 phone calls per week from the martial artist to support the training. Additionally a virtual reality device will be used to help lower stress.

SUMMARY:
The purpose of this proposed pilot study is to extend the KKC Heroes Circle program to people with opioid use disorder (OUD) who are currently enrolled in methadone maintenance treatment (MMT) and who wish to learn these techniques to reduce their behavioral and physiological dependence on medication.

The goal is to engage these MMT patients in a complementary (non-pharmacological) therapeutic activity that may improve their self-efficacy and personal control, reduce the impact of stressors and chronic pain, drug craving, affective and physical function, and lower reliance on pharmacological interventions.

DETAILED DESCRIPTION:
Overall, this project will take approximately 1 year to complete, and will be divided into three phases (each about three months long).

Phase 1: The investigators will identify and consent 10 patients, regardless of age, sex, or race/ethnicity, enrolled at the Tolan Park Research Clinic who endorse a desire to lower their daily methadone maintenance dose but have been unable to do so.

Each participant will complete a 12-week protocol. There will be twice weekly visits (each ≈30 min total for all procedures) by the trained adult Kids Kicking Cancer (KKC) martial artists. Prior to receiving his/her methadone dose, the martial artist and patient will meet in a private area to promote attention and focus on the intervention, and for measurement of biomarker data. At baseline and during weeks 4, 8 and 12, the investigators will obtain pre- and post-session saliva samples (collected with a Salivette held under the tongue 3 min) to measure two stress biomarkers. The investigators will also measure heart rate and blood pressure. Each participant will receive 20 minutes of individual instruction in a therapeutic approach to lower their stress and life challenges. Each visit will include certain martial arts rituals, including the KKC "Power, Peace, Purpose"™ mantra, and Breath Brake®, introduced by videotapes made by the "heroes" (children). Other components of the intervention session, e.g. movement exercises and mental imagery, will be tailored to the patient, always ensuring that any physical maneuver is safe for that individual. They will also receive audio meditations for smart phones or, if unavailable, loaded onto mp3 players to practice the meditations.

At the beginning and end of each visit by the martial artist, the participant will use Visual Analog Scales (VAS, 0-10 range) to rate his/her momentary level of "pain", "drug craving", "anxiety", "anger", and "depression"; and he/she will complete the short form of the Positive and Negative Affect Schedule. Each meeting will be supplemented by phone calls 3 times a week from the martial artist to each patient to supply support.

Data collection measurements: Beck Depression Inventory-II, State-Trait Anxiety Inventory, Perceived Stress Scale, Difficulties with Emotion Regulation Scale, Coping Orientation to Problems Experienced (Brief-COPE), Alcohol and Drug Use Self-Efficacy Scale, Distress Tolerance Scale, Breath-hold Endurance task, Brief Pain Inventory, Medical Outcomes Study Short Form, a computerized measure of attentional function, the Attentional Network Task, also known as Flanker Task.

Methadone dose (baseline and weekly) and urine drug test results (baseline and twice weekly for these study participants) will be extracted from the patient's medical record, with the assistance of an authorized staff member.

Each Phase I participant will undergo non-Virtual Reality (VR) intervention procedures during weeks 1-6, and will then undergo VR-based intervention during weeks 7-12.

Phase 2 will extend phase 1 by evaluating a second group of 10 patients who will also participate over a 12-week period. Identical procedures to Phase 1 will be used; in addition, the investigators will include whole-brain fMRI (functional magnetic resonance imaging) scanning before and after completion of the full intervention. Patients will use a Virtual Reality (VR) program that enables the patient to choose his/her obstacles and "see" that obstacle inside his/her head.

Phase 3 will enroll 10 additional patients (different participants from phases 1 and 2) who use opioids while complaining of specific chronic pain syndrome. In this phase, the same protocol will be used, including fMRI scanning. The Virtual Reality, however, will focus specifically on creating the image of the pain in wherever the pain is being reported in the body.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of Opioid Use Disorder
2. Stable daily methadone dose for at least one month prior to enrollment
3. Desire to reduce the daily methadone dose at least 20%.

Exclusion Criteria:

1. Pregnant (urine test) or lactating (self-report)
2. Current severe Axis I psychiatric disorder, e.g. psychosis, bipolar disorder
3. Suicidal ideation/attempt during the past year
4. Medical contraindications to the proposed therapeutic program, in the opinion of the clinic physician.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with opioid use disorder (OUD), currently enrolled in methadone maintenance treatment (MMT) who wish to learn techniques to reduce their behavioral and physiological dependence on medication.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change in methadone dose | Once at baseline and twice-weekly over a 12-week period.
  Extracted from the patient's medical record
Drug-free urine test results (<300 ng/ml) for opioids, cocaine, benzodiazepines, and barbiturates (<300 ng/ml), and cannabinoids (<50 ng/ml). | Once at baseline and twice-weekly over a 12-week period.
  Extracted from the patient's medical record

SECONDARY OUTCOMES:
Change in self-report of pain, drug craving, anxiety, anger and depression | Beginning and end of each visit by the martial artist (pre/post effects); Once at baseline and twice-weekly over a 12-week period.
  Measured by Visual Analog Scales (0: Not all all (Better outcome) - 10: Extremely (Worse outcome)
Change in self-report of the following feelings and emotions: Afraid, Ashamed, Hostile, Nervous and Upset | Beginning and end of each visit by the martial artist (pre/post effects); Once at baseline and twice-weekly over a 12-week period.
  Measured by Negative Affect Schedule (1: Very slightly or not at all (Better outcome), 2: A little, 3: Moderately, 4: Quite a bit, 5: Extremely (Worse outcome)
Change in heart rate biomarker (beats per minute (bpm) | Once at baseline and once during week 4, week 8, and week 12 over the 12-week period for a total of 4 collections.
  The investigators will obtain pre and post session heart rate measurements collected using non-invasive vital monitor
Change in blood pressure (Systolic and Diastolic mmHg) biomarker | Once at baseline and once during week 4, week 8, and week 12 over the 12-week period for a total of 4 collections.
  The investigators will obtain pre and post session blood pressure measurements collected using non-invasive vital monitor
Change in saliva cortisol biomarkers | Once at baseline and once during week 4, week 8, and week 12 over the 12-week period for a total of 4 collections.
  The investigators will obtain pre and post session saliva samples to measure saliva cortisol collected using Salivette held under tongue
Change in C-reactive protein biomarkers | Once at baseline and once during week 4, week 8, and week 12 over the 12-week period for a total of 4 collections.
  The investigators will obtain pre and post session saliva samples to measure C-reactive protein collected using Salivette held under tongue
Percentage of patients who reduce methadone dose at least 20 percent | Once at baseline and twice-weekly over a 12-week period.
  Extracted from the patient's medical record

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No